CLINICAL TRIAL: NCT02903407
Title: Pain, Agitation and Delirium Protocol in Ventilated Patients in the Duke CICU
Brief Title: Pain, Agitation and Delirium (PAD) Protocol in the Duke CICU
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: All enrolled participants completed the study protocol but the study was terminated prior to the goal number of participants due to low recruitment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00074866
Record Dates: First submitted 2016-09-02; First posted 2016-09-16 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Deep Sedation; Ventilators, Mechanical; Critical Illness
Keywords: Ventilators, Mechanical; Intensive Care Units; Deep Sedation
MeSH Terms: conditions — Critical Illness | interventions — Midazolam; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Midazolam (Active Comparator): IV midazolam will be administered for sedation while patient is mechanically ventilated. Patient will be monitored per standard of care in the CICU using the Richmond Agitation and Sedation Scale (RASS) with a set goal sedation level of RASS 0 to -2. Pain will be monitored based on the Critical-Care Pain Observation Tool (CPOT) assessment with goal less than or equal to 2. Delirium will be evaluated based on the Confusion Assessment Method for the ICU (CAM-ICU) with goal of negative or patient's baseline.
  Interventions: Drug: Midazolam
- Propofol or Dexmedetomidine (Active Comparator): Propofol or Dexmedetomidine per physician discretion will be administered for sedation while patient is mechanically ventilated. Patient will be monitored per standard of care in the CICU using the Richmond Agitation and Sedation Scale (RASS) with a set goal sedation level of RASS 0 to -2. Pain will be monitored based on the Critical-Care Pain Observation Tool (CPOT) assessment with goal less than or equal to 2. Delirium will be evaluated based on the Confusion Assessment Method for the ICU (CAM-ICU) with goal of negative or patient's baseline.
  Interventions: Drug: Propofol; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — IV midazolam will be administered as a continuous infusion to maintain set goal sedation level of RASS 0 to -2.
  Other Names: Versed
  Arms: Midazolam
Drug: Propofol — IV propofol will be administered as a continuous infusion to maintain set goal sedation level of RASS 0 to -2.
  Other Names: Diprivan
  Arms: Propofol or Dexmedetomidine
Drug: Dexmedetomidine — IV dexmedetomidine will be administered as a continuous infusion to maintain set goal sedation level of RASS 0 to -2.
  Other Names: Precedex
  Arms: Propofol or Dexmedetomidine

SUMMARY:
This study aims to examine the use of protocol directed sedation using the Duke PAD protocol with the current sedation medications of propofol or dexmedetomidine compared to the PAD protocol with midazolam, per cardiac intensive care unit (CICU) usual care, as an initial step toward understanding the best management of sedation in these patients.

DETAILED DESCRIPTION:
The optimal approach to management of sedation in the Intensive Care Unit (ICU) has become a topic of increasing interest. The most recent guidelines outline the pharmacologic mechanisms of commonly used medications as well as scales on which to measure goals of pain, sedation, agitation and delirium in the critically ill patient. This guideline is based on a cadre of randomized controlled trials examining the medications in the medical intensive care unit and post cardiac surgery patient. Notably, in each of the trials, patients presenting with acute myocardial infarction, heart failure or cardiogenic shock have been excluded or largely underrepresented.

Using the current guidelines as a foundation, a new pain, agitation and delirium (PAD) protocol, which prioritizes the use of propofol or dexmedetomidine for sedation, was developed and instituted at Duke University Hospital. However, use of this protocol in the CICU has raised important considerations. Some of these stem from the specific hemodynamic characteristics of the population, including significant bradycardia and hypotension, which can be worsened due to known side effects of propofol and dexmedetomidine. It remains unclear whether the benefits of these medications outweigh the risks in CICU patients as the use of these medications has not been studied previously in this population. This study aims to examine the use of protocol directed sedation using the Duke PAD protocol with the current sedation medications of propofol or dexmedetomidine compared to the PAD protocol with midazolam, per CICU usual care, as an initial step toward understanding the best management of sedation in these patients.

Project Aims Include:

1. Examine the efficacy of the PAD protocol using propofol or dexmedetomidine versus midazolam with regard to goal sedation, pain control and level of delirium in intubated Duke CICU patients.
2. Determine differences in duration of ventilator days, CICU stay and total hospital stay with the PAD protocol using propofol or dexmedetomidine compared to midazolam in the Duke CICU.
3. Compare the rates of adverse effects of the current PAD protocol with propofol or dexmedetomidine versus midazolam for sedation in the Duke CICU, including hypotension, bradycardia, difficulty with ventilator weaning due to sedation, and delirium.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Duke CICU, who require intubation and sedation for mechanical ventilation that is expected to be >24 hours in duration will be included, unless they meet the specified exclusion criteria.
* Patients intubated within one hour prior to care transition to the CICU will also be screened for inclusion.

Exclusion Criteria:

* Exclusion criteria include patients following resuscitation from cardiac arrest who are treated on the cooling protocol
* patients who have suffered a neurologic event (seizure, stroke) or who have baseline dementia, both of which could limit delirium assessment
* patients with child class B and C liver disease
* patients with known allergy to study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Newby, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Carson SS, Kress JP, Rodgers JE, Vinayak A, Campbell-Bright S, Levitt J, Bourdet S, Ivanova A, Henderson AG, Pohlman A, Chang L, Rich PB, Hall J. A randomized trial of intermittent lorazepam versus propofol with daily interruption in mechanically ventilated patients. Crit Care Med. 2006 May;34(5):1326-32. doi: 10.1097/01.CCM.0000215513.63207.7F. PMID 16540958
- [Background] Hall RI, Sandham D, Cardinal P, Tweeddale M, Moher D, Wang X, Anis AH; Study Investigators. Propofol vs midazolam for ICU sedation : a Canadian multicenter randomized trial. Chest. 2001 Apr;119(4):1151-9. doi: 10.1378/chest.119.4.1151. PMID 11296183
- [Background] Huey-Ling L, Chun-Che S, Jen-Jen T, Shau-Ting L, Hsing-I C. Comparison of the effect of protocol-directed sedation with propofol vs. midazolam by nurses in intensive care: efficacy, haemodynamic stability and patient satisfaction. J Clin Nurs. 2008 Jun;17(11):1510-7. doi: 10.1111/j.1365-2702.2007.02128.x. PMID 18482144
- [Background] Pandharipande PP, Sanders RD, Girard TD, McGrane S, Thompson JL, Shintani AK, Herr DL, Maze M, Ely EW; MENDS investigators. Effect of dexmedetomidine versus lorazepam on outcome in patients with sepsis: an a priori-designed analysis of the MENDS randomized controlled trial. Crit Care. 2010;14(2):R38. doi: 10.1186/cc8916. Epub 2010 Mar 16. PMID 20233428
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Searle NR, Cote S, Taillefer J, Carrier M, Gagnon L, Roy M, Lussier D. Propofol or midazolam for sedation and early extubation following cardiac surgery. Can J Anaesth. 1997 Jun;44(6):629-35. doi: 10.1007/BF03015447. PMID 9187783
- [Background] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Duke CICU between September 1, 2017 and June 30, 2019. Patients were identified by the rounding team for potential inclusion in the sedation trial and then screened by study team members to determine whether they met inclusion criteria. Consent was obtained from eligible patient's primary decision maker.
Pre-assignment Details: No enrolled participants were excluded from the study prior to group assignment.
Period: Overall Study
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Propofol or Dexmedetomidine | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72.5 [66.3 to 73.3] | 57.0 [55.5 to 63.5] | 70.0 [55.5 to 72.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 36.1 [33.2 to 38.5] | 34.4 [33.5 to 35.8] | 34.4 [33.3 to 37.7]
Ejection Fraction [Median (Inter-Quartile Range); unit: Percentage of blood] — Ejection fraction (EF) is a measurement, expressed as a percentage, of how much blood the left ventricle pumps out with each contraction.
  Percentage of blood | 30.0 [18.8 to 43.8] | 55.0 [40.0 to 55.0] | 40.0 [22.5 to 55.0]

OUTCOME MEASURES:

1. Primary Outcome: Intensive Care Unit Length of Stay
Description: Number of days of admission to the CICU during the index hospitalization
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Days | 4.1 [3.6 to 6.7] | 10.0 [8.2 to 10.3]

2. Secondary Outcome: In Hospital Mortality
Description: All-cause mortality during the hospitalization
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Number; unit: participants
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
participants | 1 | 1

3. Secondary Outcome: Hospital Length of Stay
Description: Index hospitalization length of stay in days
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Days | 19.5 [15.0 to 23.5] | 30.0 [21.5 to 35.0]

4. Secondary Outcome: Number of Participants With Increased Vasopressor Requirement
Description: Patients will be monitored for increased pressor requirement during the CICU stay
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Participants | 2 | 2

5. Secondary Outcome: Number of Participants With Bradycardia
Description: Patients will be monitored for bradycardia which may be associated with sedation drug. Average heart rate before, during and after use of drug will be recorded for each patient.
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

6. Secondary Outcome: Number of Ventilator Days
Description: Days requiring mechanical ventilation during the initial episode of intubation during the hospitalization
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Days | 2.5 [2.1 to 4.2] | 6.8 [3.9 to 8.4]

7. Secondary Outcome: Number of Days From Decision to Extubate to True Extubation
Description: The time (in days) from when the clinical care team documents a decision to pursue extubation until the time the patient was extubated
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Days | 0 [0 to 0.25] | 0 [0 to 0]

8. Secondary Outcome: Number of Days Alive During Admission and Free From Delirium or Coma
Description: The number of days alive and free from delirium or coma during admission will be evaluated among patients with CAM-ICU documented
Time Frame: One month or hospital discharge, whichever time point comes first
Population: CAM-ICU was only documented in 3/7 of the patients enrolled, all of whom were in the midazolam arm of the study. Only these patients were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 3 | 0
Days | 14.0 [13.5 to 20.0] |

9. Secondary Outcome: Percentage of Time at Goal Sedation
Description: Will use RASS (Richmond Agitation and Sedation Scale) to assess level of sedation as per standard of care by nurses in the CICU. Data that is recorded will be evaluated following discharge. The RASS ranges from -5 (unrousable) to +4 (combative) and 0 (zero) = alert and calm and goal sedation is considered a RASS level of 0 to -2.
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
percentage of time | 63.3 [43.8 to 70.8] | 63.2 [56.6 to 64.4]

10. Secondary Outcome: Time From Withdrawal of Sedation to ICU Discharge
Description: The duration, in days, from withdrawal of sedation for mechanical ventilation until the time of discharge from the ICU
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Days | 1.6 [0.77 to 2.8] | 5.6 [2.8 to 5.8]

11. Secondary Outcome: Number of Participants With Delirium
Description: Will use the Confusion Assessment Method for the ICU (CAM-ICU) to assess presence of delirium as per standard of care by nurses in the CICU. Patients with CAM-ICU data recorded will be included.
Time Frame: One month or hospital discharge, whichever time point comes first
Population: Patients with CAM-ICU score documented in the CICU (3/7 participants, all in the midazolam arm of the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 3 | 0
Participants | 1 |

12. Secondary Outcome: Pain Management
Description: Will use the CPOT (Critical-Care Pain Observation Tool) score to assess pain level as per standard of care by nurses in the CICU. The CPOT has a range of 0 to 8. A CPOT score of ≤ 2 = minimal to no pain present and >2 = unacceptable level of pain. Data that is recorded will be evaluated following discharge.
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
score on a scale | 0.0 [0.0 to 0.5] | 0.0 [0.0 to 0.3]

13. Secondary Outcome: Number of Participants Requiring Reintubation
Description: Following ICU discharge, patient charts will be reviewed to evaluate whether they required reintubation. If so, will determine whether necessity of reintubation was related to delirium.
Time Frame: One month or hospital discharge, whichever time point comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Propofol or Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From time of enrollment to hospital discharge - a range of 2-29 days for the patients enrolled in the trial
Arm/Group | Midazolam | Propofol or Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Our trial was terminated prior to goal enrollment due to difficulty with enrollment in this critically ill population of patients. The data here represent a small sample size of patients and should be viewed as pilot data for hypothesis generation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02903407/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT02903407/SAP_001.pdf